CLINICAL TRIAL: NCT05885425
Title: TELEHEART-Management of Telemedicine Monitoring of Patients With Chronic Heart Failure
Brief Title: Management of Telemedicine Monitoring of Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Trnava University in Trnava (Other)
Responsible Party: Sponsor
Other Study IDs: OPII-VA/DP/2021/9.3-01
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Congestive Heart Failure Chronic
Keywords: Congestive Heart Failure, Telemedicine
MeSH Terms: conditions — Heart Failure | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 100 patients with stabile chronic heart failure with remote control: Group 1 is the intervention group, their health status will be monitored telemetrically for a half year by several electronic devices (for measurement of hearth frequency, blood pressure, blood saturation and periodically ECG recordings). Data will be periodically transmitted to the doctor in the ambulance. If measured data will indicated any worsening of heath (decompensation of circulation), physician will adjust the treatment remotely.
  Interventions: Behavioral: Telemedicine correction of medical treatment; Behavioral: Education for proper lifestyle
- Non-intervention group: 100 patients with stabile chronic heart failure without remote control: Group 2 with patients with chronic heart failure in the non-intervention group, they will not be contacted by own physician for half a year - the planned periodic control will be scheduled after half a year.

INTERVENTIONS:
Behavioral: Telemedicine correction of medical treatment — On the basis of telemedicine data, the doctor will remotely correct medical treatment by adjusting the dose or supplementing or by omitting the medicine in order to improve the state of health, or to alleviate the symptoms of the disease monitored by telemedicine
  Groups: 100 patients with stabile chronic heart failure with remote control
Behavioral: Education for proper lifestyle — Based on telemedicine data, the doctor can consider periodic education of the patient with the innervated group in order to improve lifestyle
  Groups: 100 patients with stabile chronic heart failure with remote control

SUMMARY:
Objective: to evaluate the possibilities and effect of telemedicine monitoring and management of patients with CHF (compared to patients with CHF without intensive telemedicine monitoring) on quality of life, prognosis and the presence of complications and hospitalisations.

Patients with a stable form of congestive heart failure will be gradually included in the study. Half of them will be defined by random selection to intervention group. Parameters, that can be measured at home will be periodically telemedical monitored. In according with at home monitored data, the own physician will be able to intervene with change of medical treatment in the case of non-physiological deviations in order to improve the health status as well as the prognosis of the patient with CHF.

DETAILED DESCRIPTION:
Inclusion criteria:

* Age between 45 and 75
* Congestive heart failure (CHF), NYHA II - VI (any genesis)
* EF less then 45%, any rhythm (sinus or atrial fibrillation)
* More as two months stable condition
* Complete treatment according to recommendations (guidelines): ACEI (alternatively ARNI / sartan) + diuretics + betablockers (as alternative digitalis)
* Without hospitalization with CHF decompensation more as two months before enrolment
* No severe liver disease and hemodialysis treatment
* No planned any cardio-surgery intervention in the next six months
* No a serious valvular defects

Input and output surveys (measurements, tests) upon enrollment and after half a year ECHOCG (mandatory parameters: EF, LVDd, IVCT, E/A, LA diameter, LA area planimetrically) Blod pressure, frequency, ECG (PQ, QT, description: blockages, STT segment changes) Six minutes walking test Serum analysis: NTproBNP, CRP, natrium, potassium, urea, creatinine

Questionnaires:

* Kansas Quality of Life Questionnaire (KCCQ)
* Questionnaire SF 36 (perception of illness)
* Beck's Depression Inventory (21 questions) - depression questionnaire
* Beck's Anxiety Inventory (21 questions) - anxiety questionnaire (standardized questionnaires translated into Slovak)

Telemedicine monitoring: the patient will have at home devices for:

ECG recording Blood pressure and pulse sensor O2 saturation sensor Personal weight machine

Data will be transferred via smartphone software (supplied by the organizer) once a week too physician:

ECG recording on the patient's instructions

1. st morning in bed after waking up (stick electrodes for whole day)
2. nd. after breakfast (or an hour after getting out of bed)
3. th. around 12 o'clock (time of lunch)

In the same day morning, weight and other measurements (O2, blood pressure, pulse)

As part of the data transfer, the information for physician:

possibility to send a comment "how I feel" the number of urinations per night Data is entered into a standard table in the doctor's software (supplied by the organizer) Based on the obtained data, the doctor can correct the treatment at any time by telephone

Physician will control the transferred data from patient at least once every week.

The organizer will deliver Personal weight machine (new uniform) Questionnaires (in printed form) Informed consents devices for monitoring of physiological functions (ECG, O2, pulse, blood pressure) Application for the patient's smartphone (for simple data transfer) Software recording data from the patient to the PC at the physician's office Compensation 100,- € (motivation for each participant - intervened or non-intervened) similar compensation is assumed at the end of follow-up (for each patient) The ECG sensor will remain available to the physicians Included doctors will be co-authors of publications in foreign journals.

Monitored events ("end points"):

hospitalization for cardiac causes visit to the emergency room (urgent) calling Quick Medical Assistance at home unplanned visit by cardiologist / internist fundamental change of treatment (new type of drug, change of drug group, increased dose) fundamental changes (deterioration) in the perception of the disease (SF 36) major changes in quality of life (Kansas Questionnaire) fundamental changes in the perception of depression (Beck's Depression Inventory) fundamental changes in the perception of anxiety (Beck's Anxiety Inventory) Death

Evaluation in addition to endpoints:

long-term trend of resting frequency long-term trend of increased frequency after morning exercise and during the day long-term blood pressure and saturation trends number of telephone contacts by physicians with the patient in the case of using a "smart watch", also trends in sleep parameters (frequency, apnea, sleep quality, caloric expenditure / day)

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure (CHF), NYHA II - VI (any genesis)
* EF less then 45%, any rhythm (sinus or atrial fibrillation)
* More as two months stable condition
* Complete treatment according to recommendations (guidelines): ACEI (alternatively ARNI / sartan) + diuretics + betablockers (as alternative digitalis)
* Without hospitalization with CHF decompensation more as two months before enrolment

Exclusion Criteria:

* malignant diseases
* planned cardiac surgery

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with congestive heart failure with ejection fraction less than 45%
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for cardiac reasons | 6 months
Visit to the emergency room (urgent) | 6 months

SECONDARY OUTCOMES:
Unplanned visit to cardiology / internist | 6 months
Calling Quick Medical Assistance home | 6 months
Fundamental change of treatment (new type of drug, change of drug group, increased dose) | 6 months
Fundamental changes in the quality of life according to questionnaires | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva Goncalvesova, Principal Investigator — National Institute of Vascular and Heart Diseases Bratislava; Fedor Lehocki, Study Chair — Slovak University of Technology in Bratislava; Jozef Benacka, Study Director — Trnava University in Trnava

IPD SHARING:
Plan to Share IPD: No
No.